CLINICAL TRIAL: NCT00383708
Title: Phase III, Multicentre, Open Study to Assess the Efficacy and Safety Profiles of the Co-administration of Lanreotide Autogel 120 mg (Administered Via Deep Subcutaneous Injections Every 28 Days) and Pegvisomant 40 to 120 mg Per Week (Administered Via Subcutaneous Route Once or Twice a Week) in Acromegalic Patients Failing to Respond to Lanreotide Autogel 120 mg Alone
Brief Title: Lanreotide Autogel and Pegvisomant Combination Therapy in Acromegalic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2-55-52030-727
Record Dates: First submitted 2006-10-02; First posted 2006-10-03 (Estimated); Results first posted 2018-07-23 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — lanreotide; pegvisomant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: lanreotide (Autogel formulation); Drug: Pegvisomant

INTERVENTIONS:
Drug: lanreotide (Autogel formulation) — 120 mg administered via deep subcutaneous injection every 28 days over 28 weeks.
Drug: Pegvisomant — Administered at 40 to 120 mg per week via subcutaneous injection once or twice a week over 28 weeks.

SUMMARY:
The main aim of this study is to assess the efficacy of the co-administration of lanreotide Autogel 120 mg (administered via deep sub-cutaneous injections every 28 days) and pegvisomant (administered at 40 to 120 mg per week via sub-cutaneous injection given once or twice a week) on IGF-1 levels over 28 weeks in acromegalic patients. The primary endpoint will be the percentage of acromegalic patients with normalised (age and sex adjusted) IGF-1 level at the end of the co-treatment period.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have had documentation supporting the diagnosis of acromegaly, including elevated GH and/or IGF-1 levels
* The patient is treated with pegvisomant, because of IGF-1 level remaining above ULN when treated with somatostatin analogue, on a daily basis for at least 3 months and has normal (age and sex adjusted) IGF-1 level, or IGF-1 level above the upper limit of normal (ULN) after treatment with pegvisomant 30 mg per day, OR the patient is treated with lanreotide Autogel or octreotide LAR for at least 6 months including 3 months at the highest marketed dose and has a serum IGF-1 level above ULN, 28 days after the last injection
* At the end of the run-in period, The patient has a serum IGF-1 level above 1.2 x ULN, or a serum IGF-1 level between ULN and 1.2 x ULN and a serum GH nadir > 1 µg/L (assessed by an OGTT), 28 days after the 3rd injection of lanreotide Autogel 120 mg OR the patient is diabetic and has a serum IGF-1 level above 1.2 ULN, 28 days after the 3rd injection of lanreotide Autogel 120 mg

Exclusion Criteria:

* The patient has undergone pituitary surgery or radiotherapy within 6 months prior to study entry, or it is anticipated that it will be done during the study
* The patient has already been treated with a somatostatin analogue associated with a GH antagonist
* The patient has received dopamine agonist within 6 weeks prior to the study entry
* The patient has abnormal hepatic function at study entry (defined as AST, ALT, GGT, alkaline phosphatase, prothrombin time or total bilirubin above 2 ULN)
* The patient is at risk of pregnancy or is lactating

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2006-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (24):
- Czechia (2):
  - University Hospital, Charles University, Hradec Králové
  - Charles University, Prague
- Aarhus Kommunehospital, Aarhus, Denmark
- France (5):
  - Groupe Hospitalier Henri Mondor- Albert Chenevier, Créteil
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Clinique Marc Linquette, Lille
  - Hôpital de la Timone, Marseille
  - CHU de Rangueil, Toulouse
- Germany (3):
  - Charite Campus Mitte, Berlin
  - Klinikum Johann Wolfgang Goethe-Universität, Frankfurt
  - Medizinische Klinik Innenstadt, München
- Anticancer Hospital Metaxa Piraeus, Piraeus, Greece
- Italy (3):
  - Universitá degli Studi di Milano, Milan
  - University Federico II, Napoli
  - Universitá di Torino, Torino
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Dept. of Internal Medicine Erasmus MC, Rotterdam
- Spain (3):
  - Hospital General de Alicante, Alicante
  - Clínica Puerta de Hierro, Madrid
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Uppsala University Hospital, Uppsala
- United Kingdom (2):
  - Christie Hospital and Holt Radium Institute, Manchester
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers/

REFERENCES:
- [Result] van der Lely AJ, Bernabeu I, Cap J, Caron P, Colao A, Marek J, Neggers S, Birman P. Coadministration of lanreotide Autogel and pegvisomant normalizes IGF1 levels and is well tolerated in patients with acromegaly partially controlled by somatostatin analogs alone. Eur J Endocrinol. 2011 Mar;164(3):325-33. doi: 10.1530/EJE-10-0867. Epub 2010 Dec 10. PMID 21148630

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was a multicentre, open, single arm, sequential study where subjects were recruited to 25 study centres across 10 European countries. Subjects were enrolled to the study from 02 October 2006 (first subject enrolled) until 27 October 2008 (last subject completed).
Pre-assignment Details: A total of 125 patients were screened. Subjects were assigned to treatment if they met all inclusion and none of the exclusion criteria. 92 subjects received treatment during the run-in period and 57 subjects received treatment during the co-administration period.
Groups:
- All Subjects: Subjects confirmed as eligible for the study were entered into a run-in period of 16 weeks during which they received one deep subcutaneous (s.c.) injection of lanreotide Autogel 120 mg every 28 days. If after completion of the run-in period, subjects met the eligibility criteria for levels of serum IGF-1 (and serum growth hormone [GH] nadir), they were entered into the co-administration period during which they received both lanreotide Autogel and pegvisomant concomitantly for 28 weeks. The lanreotide Autogel dose during the co-administration period was fixed at 120 mg. Pegvisomant was administered once or twice a week via s.c. injection and the dose of could be adapted every 8 weeks based on insulin-like growth factor 1 (IGF-1) levels, following a starting dose of 60 mg once a week (dose could vary from 40 to 120 mg per week and maximum permitted dose was 60 mg twice a week).
Period: Enrolment Through Start Treatment
Arm/Group | All Subjects
Started | 125
Completed | 92
Not Completed | 33
Not completed — Withdrawal by Subject | 1
Not completed — Did not meet entry criteria | 32
Period: Run-in Period
Arm/Group | All Subjects
Started | 92
Completed | 85
Not Completed | 7
Not completed — Protocol Violation | 4
Not completed — Adverse Event | 2
Not completed — Claustrophobia | 1
Period: Co-administration Period
Arm/Group | All Subjects
Started (28 subjects were not eligible for co-administration period based on IGF-1 levels and were withdrawn) | 57
Completed | 52
Not Completed | 5
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the intention to treat (ITT) population which was defined as all co-administered subjects (i.e. treated with at least one dose of each of the two IMPs within the co-administration period) having at least one baseline and at least one post-baseline assessment of the primary efficacy endpoint.
Groups:
- Lanreotide Autogel + Pegvisomant Co-administration: Eligible subjects were entered into the co-administration period during which they received both lanreotide Autogel and pegvisomant concomitantly for 28 weeks. The lanreotide Autogel dose during the co-administration period was fixed at 120 mg and was administered by one deep s.c. injection every 28 days. Pegvisomant was administered once or twice a week via s.c. injection. The starting dose was 60 mg once a week dose. Dose adaptation of pegvisomant could then be made every 8 weeks based on IGF-1 levels taken 4 weeks after previous dose adaptation and by the third titration, subjects could receive either 40 mg, 60 mg or 80 mg once a week or 40 mg or 60 mg twice per week.
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Acromegaly With a Normalised (Age and Sex Adjusted) IGF-1 Level at the End of the Co-administration Period
Description: Serum IGF-1 is a well known and validated marker of acromegaly. IGF-1 assessments were performed at Visit (V) 1, V2, V3, V5, V7, V9 and V11 (or in case of premature study discontinuation, at the early withdrawal visit) and were based on a single serum sample taken in fasting conditions, prior to investigational medicinal product (IMP) administration. Percentage of subjects with a normalised (age and sex adjusted) IGF-1 level at the end of the co-administration period are presented. The last observation carried forward (LOCF) was used to replace missing IGF-1 values.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: The ITT population was defined as all co-administered subjects (treated with at least one dose of each of the two IMPs within the co-administration period) having at least one baseline and at least one post-baseline assessment of the primary efficacy endpoint.
Measure: Number; unit: percentage of subjects
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
percentage of subjects | 57.9
Statistical Analysis 1: Comparison: Lanreotide Autogel + Pegvisomant Co-administration; The percentage of subjects (denoted as pnor) was compared to the minimum clinically relevant (theoretical) percentage of 30%, using an exact test based on the binomial distribution. The test was an upper-tailed test of H0: pnor ≤ 0.3 versus H1: pnor > 0.3; Test type: Other; p < 0.0001, Exact test; One-sided p value

2. Primary Outcome: Percentage of Subjects With Acromegaly With a Normalised (Age and Sex Adjusted) IGF-1 Level at the End of the Co-administration Period; Summarised by Previous Treatment and by Final Dose of Pegvisomant
Description: Serum IGF-1 is a well known and validated marker of acromegaly. IGF-1 assessments were performed at V1, V2, V3, V5, V7, V9 and V11 (or in case of premature study discontinuation, at the early withdrawal visit) and were based on a single serum sample taken in fasting conditions, prior to IMP administration. Percentage of subjects with a normalised (age and sex adjusted) IGF-1 level at the end of the co-administration period, summarised by previous treatment and by final pegvisomant dose are presented. The denominator used to calculate percentages was the number of subjects in each subgroup, comprising previous treatment with pegvisomant, lanreotide Autogel and octreotide long acting repeatable (LAR) and final pegvisomant dose as either 40 mg, 60 mg or 80 mg once a week or 40 mg or 60 mg twice per week. The LOCF approach was used to replace missing IGF-1 values.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: The ITT population was defined as all co-administered subjects (treated with at least one dose of each of the two IMPs within the co-administration period) having at least one baseline and at least one post-baseline assessment of the primary efficacy endpoint. Only evaluable subjects within each individual subgroup analysed for each category.
Measure: Number; unit: percentage of subjects
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
percentage of subjects
  Previous Treatment: Pegvisomant: number analyzed (Participants) | 13
  Previous Treatment: Pegvisomant | 46.2
  Previous Treatment: Lanreotide Autogel: number analyzed (Participants) | 24
  Previous Treatment: Lanreotide Autogel | 54.2
  Previous Treatment: Octreotide LAR: number analyzed (Participants) | 20
  Previous Treatment: Octreotide LAR | 70.0
  Final Dose Pegvisomant: 40 mg/week: number analyzed (Participants) | 13
  Final Dose Pegvisomant: 40 mg/week | 76.9
  Final Dose Pegvisomant: 60 mg/week: number analyzed (Participants) | 13
  Final Dose Pegvisomant: 60 mg/week | 61.5
  Final Dose Pegvisomant: 80 mg/week: number analyzed (Participants) | 16
  Final Dose Pegvisomant: 80 mg/week | 75.0
  Final Dose Pegvisomant: 40 mg 2x/week: number analyzed (Participants) | 5
  Final Dose Pegvisomant: 40 mg 2x/week | 60.0
  Final Dose Pegvisomant: 60 mg 2x/week: number analyzed (Participants) | 10
  Final Dose Pegvisomant: 60 mg 2x/week | 0
Statistical Analysis 1: Comparison: Lanreotide Autogel + Pegvisomant Co-administration; The percentage of subjects in the subgroup previously treated with pegvisomant (denoted as pnor) was compared to the minimum clinically relevant (theoretical) percentage of 30%, using an exact test based on the binomial distribution. The test was an upper-tailed test of H0: pnor ≤ 0.3 versus H1: pnor > 0.3; Test type: Other; p = 0.1654, Exact test — One-sided p value
Statistical Analysis 2: Comparison: Lanreotide Autogel + Pegvisomant Co-administration; The percentage of subjects in the subgroup previously treated with lanreotide Autogel (denoted as pnor) was compared to the minimum clinically relevant (theoretical) percentage of 30%, using an exact test based on the binomial distribution. The test was an upper-tailed test of H0: pnor ≤ 0.3 versus H1: pnor > 0.3; Test type: Other; p = 0.0115, Exact test — One-sided p value
Statistical Analysis 3: Comparison: Lanreotide Autogel + Pegvisomant Co-administration; The percentage of subjects in the subgroup previously treated with octreotide LAR (denoted as pnor) was compared to the minimum clinically relevant (theoretical) percentage of 30%, using an exact test based on the binomial distribution. The test was an upper-tailed test of H0: pnor ≤ 0.3 versus H1: pnor > 0.3; Test type: Other; p = 0.0003, Exact test — One-sided p value

3. Primary Outcome: Percentage of Subjects With Acromegaly With a Normalised (Age and Sex Adjusted) IGF-1 Level at the End of the Co-administration Period; Summarised by Diabetic Status at Baseline
Description: Serum IGF-1 is a well known and validated marker of acromegaly. IGF-1 assessments were performed at V1, V2, V3, V5, V7, V9 and V11 (or in case of premature study discontinuation, at the early withdrawal visit) and were based on a single serum sample taken in fasting conditions, prior to IMP administration. Percentage of subjects with a normalised (age and sex adjusted) IGF-1 level at the end of the co-administration period, summarised by diabetic status are presented. The denominator used to calculate percentages was the number of subjects in each subgroup (diabetic and non diabetic). The LOCF approach was used to replace missing IGF-1 values.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: The ITT population was defined as all co-administered subjects (treated with at least one dose of each of the two IMPs within the co-administration period) having at least one baseline and at least one post-baseline assessment of the primary efficacy endpoint. Only evaluable subjects within each of the two subgroups analysed for each category.
Measure: Number; unit: percentage of subjects
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
percentage of subjects
  Diabetic Subjects: number analyzed (Participants) | 19
  Diabetic Subjects | 47.4
  Non Diabetic Subjects: number analyzed (Participants) | 38
  Non Diabetic Subjects | 63.2
Statistical Analysis 1: Comparison: Lanreotide Autogel + Pegvisomant Co-administration; The percentage of subjects in the subgroup diabetic subjects (denoted as pnor) was compared to the minimum clinically relevant (theoretical) percentage of 30%, using an exact test based on the binomial distribution. The test was an upper-tailed test of H0: pnor ≤ 0.3 versus H1: pnor > 0.3; Test type: Other; p = 0.084, Exact test — One-sided p value
Statistical Analysis 2: Comparison: Lanreotide Autogel + Pegvisomant Co-administration; The percentage of subjects in the subgroup non diabetic subjects (denoted as pnor) was compared to the minimum clinically relevant (theoretical) percentage of 30%, using an exact test based on the binomial distribution. The test was an upper-tailed test of H0: pnor ≤ 0.3 versus H1: pnor > 0.3; Test type: Other; p < 0.0001, Exact test — One-sided p value

4. Secondary Outcome: Percentage of Subjects With a Normalised (Age and Sex Adjusted) IGF-1 Level at Any Time During the Co-administration Period
Description: Serum IGF-1 is a well known and validated marker of acromegaly. IGF-1 assessments were performed at V1, V2, V3, V5, V7, V9 and V11 (or in case of premature study discontinuation, at the early withdrawal visit) and were based on a single serum sample taken in fasting conditions, prior to IMP administration. Percentage of subjects with a normalised (age and sex adjusted) IGF-1 level at least once during the co-administration period, summarised by 'while taking the final dose during co-administration' and 'at any time during co-administration' are presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
percentage of subjects
  While Taking Final Dose During Co-administration | 66.7
  At Any Time During Co-administration | 78.9
Statistical Analysis 1: Comparison: Lanreotide Autogel + Pegvisomant Co-administration; The percentage of subjects in the subgroup 'while taking final dose during co-administration' (denoted as pnor) was compared to the minimum clinically relevant (theoretical) percentage of 30%, using an exact test based on the binomial distribution. The test was an upper-tailed test of H0: pnor ≤ 0.3 versus H1: pnor > 0.3; Test type: Other; p < 0.0001, Exact test — One-sided p-value
Statistical Analysis 2: Comparison: Lanreotide Autogel + Pegvisomant Co-administration; The percentage of subjects in the subgroup 'at any time during co-administration' (denoted as pnor) was compared to the minimum clinically relevant (theoretical) percentage of 30%, using an exact test based on the binomial distribution. The test was an upper-tailed test of H0: pnor ≤ 0.3 versus H1: pnor > 0.3; Test type: Other; p < 0.0001, Exact test — One-sided p-value

5. Secondary Outcome: Percentage of Subjects With Normalised (Age and Sex Adjusted) IGF-1 at Each Assessment
Description: Serum IGF-1 is a well known and validated marker of acromegaly. IGF-1 assessments were performed at V1, V2, V3, V5, V7, V9 and V11 (or in case of premature study discontinuation, at the early withdrawal visit) and were based on a single serum sample taken in fasting conditions, prior to IMP administration. The percentage of subjects with a normalised (age and sex adjusted) IGF-1 level is presented. The denominator used to calculate the percentages was the number of ITT population subjects with an assessment at the visit. In addition to the data for each individual visit, the last value available (LVA) data is also presented. None of the ITT population subjects had serum IGF-1 normalised at V3, consistent with the criterion to continue in the study and be treated in the co-administration period.
Time Frame: V1 (Screening) up to V11 (Week 44)
Population: The ITT population was defined as all co-administered subjects (treated with at least one dose of each of the two IMPs within the co-administration period) having at least one baseline and at least one post-baseline assessment of the primary efficacy endpoint. Only evaluable subjects with assessments at each specified visit included in analysis.
Measure: Number; unit: percentage of subjects
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
percentage of subjects
  V1 (Screening) | 17.5
  V2 (Day 1): number analyzed (Participants) | 53
  V2 (Day 1) | 24.5
  V3 (Week 12): number analyzed (Participants) | 0
  V5 (Week 20): number analyzed (Participants) | 55
  V5 (Week 20) | 56.4
  V7 (Week 28): number analyzed (Participants) | 54
  V7 (Week 28) | 48.1
  V9 (Week 36): number analyzed (Participants) | 52
  V9 (Week 36) | 57.7
  V11 (Week 44): number analyzed (Participants) | 52
  V11 (Week 44) | 61.5
  LVA | 57.9

6. Secondary Outcome: Change From Baseline in Serum IGF-1 Levels (Expressed as Z-scores) During the Co-administration Period
Description: The change in serum IGF-1 levels, expressed as z-scores calculated using the age and sex specific mean and standard deviation [SD] values from Baseline to V11 and to LVA are presented. A z-score between +/- 2 indicates a normal IGF-1 concentration.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
z-score
  Change at V11: number analyzed (Participants) | 52
  Change at V11 | -4.50 (4.01)
  Change at LVA | -4.25 (4.00)

7. Secondary Outcome: Change From Baseline in Acromegaly Symptoms During the Co-administration Period
Description: Acromegaly symptoms, including arthralgia, excessive perspiration, fatigue, headache and soft tissue swelling were assessed with scores ranging from 0 (no symptoms) to 8 (severe, incapacitating symptoms). Symptoms were assessed by the subject in paper format before any other procedure planned during the visit. The change in acromegaly symptoms from Baseline to V11 and to LVA are presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 56
units on a scale
  Arthralgia: Change at V11: number analyzed (Participants) | 50
  Arthralgia: Change at V11 | -0.7 (1.5)
  Arthralgia: Change at LVA | -0.6 (1.6)
  Excessive Perspiration: Change at V11: number analyzed (Participants) | 50
  Excessive Perspiration: Change at V11 | -0.4 (1.9)
  Excessive Perspiration: Change at LVA | -0.4 (1.8)
  Fatigue: Change at V11: number analyzed (Participants) | 50
  Fatigue: Change at V11 | -0.2 (1.6)
  Fatigue: Change at LVA | -0.2 (1.5)
  Headache: Change at V11: number analyzed (Participants) | 49
  Headache: Change at V11 | -0.4 (1.6)
  Headache: Change at LVA: number analyzed (Participants) | 55
  Headache: Change at LVA | -0.3 (1.6)
  Soft Tissue Swelling: Change at V11: number analyzed (Participants) | 50
  Soft Tissue Swelling: Change at V11 | -0.6 (1.9)
  Soft Tissue Swelling: Change at LVA | -0.6 (1.8)

8. Secondary Outcome: Change From Baseline in Acromegaly Quality of Life (ACROQoL) Assessments During the Co-administration Period
Description: The ACROQoL is a health-related quality of life (QoL) questionnaire for patients with acromegaly consisting of 22 items measured on a 5-point Likert-type scale that assesses frequency of occurrence (always to never) or degree of agreement (completely agree to completely disagree) with the statements. The ACROQoL consists of questions that evaluate physical (8 items) and psychological aspects related to appearance and personal relations (7 items each). Answers are transformed to a percentage value, where 100 is the maximal (best) and 0 the minimum (worse) score depicting self-perceived quality QoL. An increase in ACROQoL score is associated with an improved QoL. The change in ACROQoL global score, physical and psychological dimension scores and appearance and personal relationships sub-dimension scores from Baseline to V11 and to LVA are presented. Relnship = Relationship; Dim = Dimension.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
units on a scale
  Global Score: Change at V11: number analyzed (Participants) | 52
  Global Score: Change at V11 | 2.4 (9.1)
  Global Score: Change at LVA | 2.2 (8.8)
  Physical Dimensions Score: Change at V11: number analyzed (Participants) | 52
  Physical Dimensions Score: Change at V11 | 4.2 (12.0)
  Physical Dimensions Score: Change at LVA | 3.5 (12.0)
  Psychological Dimensions Score: Change at V11: number analyzed (Participants) | 52
  Psychological Dimensions Score: Change at V11 | 1.3 (10.4)
  Psychological Dimensions Score: Change at LVA | 1.4 (10.0)
  Appearance Sub-Dimension Score: Change at V11 | 3.8 (13.0)
  Appearance Sub-Dimension Score: Change at LVA: number analyzed (Participants) | 52
  Appearance Sub-Dimension Score: Change at LVA | 3.7 (12.4)
  Personal Relnship Sub-Dim Score: Change at V11: number analyzed (Participants) | 52
  Personal Relnship Sub-Dim Score: Change at V11 | -0.1 (12.7)
  Personal Relnship Sub-Dim Score: Change at LVA | -0.9 (12.2)

9. Secondary Outcome: Correlation Between the Changes in ACROQoL Assessments With the Corresponding Changes in Z-score of IGF-1 Levels Over the Run-in Period and Co-administration Period
Description: The correlation between the changes in ACROQoL (expressed as standardised scores and undertaken for global score, physical and psychological dimension scores and appearance and personal relationships sub-dimension scores) over the run-in period (V3 minus V2) and co-administration period (V11 and LVA minus V3) with the corresponding changes in z-score for the IGF-1 level is presented. A decrease in IGF-1 z-score represents an improvement and an increase in ACROQoL score represents an improvement. Spearman's rank correlation (r) values are presented for change from V2 to V3 (Baseline) and from Baseline to V11/LVA for each of the specified ACROQoL categories. Corr = Correlation; Dim = Dimension; Relnship = Relationship.
Time Frame: At V2 (Day 1; Run-in), V3 (Week 12; Baseline) and V11 (Week 44)
Population: as for outcome 1
Measure: Number; unit: correlation value
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
correlation value
  Corr: Change V2 to V3 for Global Score | -0.16
  Corr: Change V3 to V11/LVA for Global Score | 0.09
  Corr: Change V2 to V3 for Physical Dim | -0.17
  Corr: Change V3 to V11/LVA for Physical Dim | 0.14
  Corr: Change V2 to V3 for Psychological Dim | -0.1
  Corr: Change V3 to V11/LVA for Psychological Dim | 0.08
  Corr: Change V2 to V3 for Appearance | -0.12
  Corr: Change V3 to V11/LVA for Appearance | 0.04
  Corr: Change V2 to V3 for Personal Relnship | -0.01
  Corr: Change V3 to V11/LVA; Personal Relnship | 0.02

10. Other Pre Specified Outcome: Change From Baseline in Serum GH Levels During the Co-administration Period
Description: Serum samples were assessed for GH levels at the same timepoints as the IGF-1 sample at V1 and V2 and during the OGTT (non diabetic subjects only) at V3 and V11 (or at the early withdrawal visit in case of premature discontinuation). Five samples were taken over 2 hours in order to assess GH nadir and confirm the subject's eligibility before entering the co-administration period. For diabetic subjects, the OGTT was replaced by a measurement of GH level on a blood sample taken at the same time as IGF-1 at V3 and V11 (or at the early withdrawal visit). The change in mean serum GH levels from Baseline to V11 and to LVA is presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
nanograms per millilitre (ng/mL)
  Change at V11: number analyzed (Participants) | 52
  Change at V11 | 6.6 (9.9)
  Change at LVA | 6.6 (9.7)

11. Other Pre Specified Outcome: Percentage of Subjects With Serum GH Levels Lesser or Equal to 2.5 ng/mL During the Study
Description: Serum samples were assessed for GH levels at the same timepoints as the IGF-1 sample at V1 and V2 and during the OGTT (non diabetic subjects only) at V3 and V11 (or at the early withdrawal visit in case of premature discontinuation). Five samples were taken over 2 hours in order to assess GH nadir and confirm the subject's eligibility before entering the co-administration period. For diabetic subjects, the OGTT was replaced by a measurement of GH level on a blood sample taken at the same time as IGF-1 at V3 and V11 (or at the early withdrawal visit). The percentage of subjects with serum GH levels ≤ 2.5 ng/mL at Baseline, V11 and LVA is presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
percentage of subjects
  At V3 | 38.6
  At V11: number analyzed (Participants) | 52
  At V11 | 25.0
  At LVA | 22.8

12. Other Pre Specified Outcome: Change From Baseline in Serum GH Binding Protein Levels During the Co-administration Period
Description: Serum samples were assessed for GH binding protein levels at V1, V2, V3 and V11 (or at the early withdrawal visit in case of premature discontinuation). The change in mean serum GH binding protein from Baseline to V11 and to LVA is presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
pmol/L
  Change at V11: number analyzed (Participants) | 52
  Change at V11 | 841 (302)
  Change at LVA | 811 (320)

13. Other Pre Specified Outcome: Change From Baseline in Acid Labile Subunit Levels From Baseline During the Co-administration Period
Description: Serum samples were assessed for acid labile subunit levels at V1, V2, V3 and V11 (or at the early withdrawal visit in case of premature discontinuation). The change in mean acid labile subunit levels from Baseline to V11 and to LVA is presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: milli IU per millilitre (mIU/mL)
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
milli IU per millilitre (mIU/mL)
  Change at V11: number analyzed (Participants) | 52
  Change at V11 | -561 (528)
  Change at LVA | -541 (522)

14. Other Pre Specified Outcome: Change From Baseline in Prolactin Levels During the Co-administration Period
Description: Serum samples were assessed for prolactin levels at V1, V2, V3 and V11 (or at the early withdrawal visit in case of premature discontinuation). The change in mean prolactin levels from Baseline to V11 and to LVA is presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: micrograms per litre (mcg/L)
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
micrograms per litre (mcg/L)
  Change at V11: number analyzed (Participants) | 52
  Change at V11 | -0.1 (8.9)
  Change at LVA | -0.4 (8.8)

15. Secondary Outcome: Change From Baseline in Mean Weight From Baseline During the Co-administration Period
Description: Weight was recorded at V2, V3 and V11 (or in case of premature study discontinuation, at the early withdrawal visit). The change in mean weight from Baseline to V11 and to LVA are presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: The Safety population was defined as all subjects who received at least one dose of each IMP during the co-administration period (i.e. one dose of lanreotide Autogel 120 mg and one dose of pegvisomant). Only evaluable subjects with an assessment at the specified visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 53
kilograms (kg)
  Change at V11: number analyzed (Participants) | 49
  Change at V11 | -0.3 (2.9)
  Change at LVA | -0.3 (2.9)

16. Secondary Outcome: Change From Baseline in Mean Supine Systolic and Diastolic Blood Pressure (BP) During the Co-administration Period
Description: Blood pressure (supine after resting for 3 minutes) was recorded at V1, V2, V3, V5, V7, V9 and V11 (or in case of premature study discontinuation, at the early withdrawal visit). The change in mean BP (systolic and diastolic) from Baseline to V11 and to LVA are presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: millimetres mercury (mmHg)
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
millimetres mercury (mmHg)
  Supine Systolic BP: Change at V11: number analyzed (Participants) | 52
  Supine Systolic BP: Change at V11 | -0.4 (17.1)
  Supine Systolic BP: Change at LVA | 0.2 (16.6)
  Supine Diastolic BP: Change at V11: number analyzed (Participants) | 52
  Supine Diastolic BP: Change at V11 | -0.1 (11.4)
  Supine Diastolic BP: Change at LVA | -0.3 (11.5)

17. Secondary Outcome: Change From Baseline in Mean Supine Heart Rate During the Co-administration Period
Description: Heart rate (supine after resting for 3 minutes) was recorded at V1, V2, V3, V5, V7, V9 and V11 (or in case of premature study discontinuation, at the early withdrawal visit). The change in mean heart rate from Baseline to V11 and to LVA are presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
beats per minute (bpm)
  Change at V11: number analyzed (Participants) | 50
  Change at V11 | -3.1 (12.6)
  Change at LVA | -2.5 (12.7)

18. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG) Mean Heart Rate During the Co-administration Period
Description: Twelve-lead ECG recordings were performed at V2, V3 and V11. Sinus rhythm, heart rate, PR interval, RR interval, QRS interval and QT interval were measured and heart rate corrected QT interval using the Fridericia method (QTcF) was calculated. The change in ECG mean heart rate from Baseline to V11 and to LVA is presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: The Safety population was defined as all subjects who received at least one dose of IMP drug during the co-administration period (i.e. one dose of lanreotide Autogel 120 mg and one dose of pegvisomant). Only evaluable subjects with an assessment at the specified visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 53
bpm
  Change at V11: number analyzed (Participants) | 50
  Change at V11 | -2.8 (11.0)
  Change at LVA | -2.2 (11.2)

19. Secondary Outcome: Change From Baseline in Mean PR Interval, QRS Interval, QT Interval, RR Interval and QTcF During the Co-administration Period
Description: Twelve-lead ECG recordings were performed at V2, V3 and V11. Sinus rhythm, heart rate, PR interval, RR interval, QRS interval and QT interval were measured and QTcF was calculated. The change in mean ECG parameter for PR interval, QRS interval, QT interval, RR interval and QTcF from Baseline to V11 and to LVA are presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: The Safety population was defined as all subjects who received at least one dose of each IMP during the co-administration period (i.e. one dose of lanreotide Autogel 120 mg and one dose of pegvisomant). Only evaluable subjects with an assessment at the specified visit were included in each individual analysis.
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 53
milliseconds (ms)
  PR Interval: Change at V11: number analyzed (Participants) | 48
  PR Interval: Change at V11 | 1.1 (15.8)
  PR Interval: Change at LVA: number analyzed (Participants) | 51
  PR Interval: Change at LVA | 1.3 (15.5)
  QRS Interval: Change at V11: number analyzed (Participants) | 50
  QRS Interval: Change at V11 | 0.1 (10.1)
  QRS Interval: Change at LVA | 0.3 (10.1)
  QT Interval: Change at V11: number analyzed (Participants) | 45
  QT Interval: Change at V11 | 4.0 (29.7)
  QT Interval: Change at LVA: number analyzed (Participants) | 48
  QT Interval: Change at LVA | 2.4 (29.9)
  RR Interval: Change at V11: number analyzed (Participants) | 50
  RR Interval: Change at V11 | 34.7 (175.4)
  RR Interval: Change at LVA | 27.6 (174.8)
  QTcF: Change at V11: number analyzed (Participants) | 45
  QTcF: Change at V11 | -1.8 (16.9)
  QTcF: Change at LVA: number analyzed (Participants) | 48
  QTcF: Change at LVA | -2.2 (16.6)

20. Secondary Outcome: Number of Subjects With Shift in Presence/Absence of Lithiasis and/or Sludge During Co-administration Period
Description: A gallbladder ultrasound was performed at V2, V3, and V11 (or in case of premature study discontinuation, at the early withdrawal visit). Presence of lithiasis and sludge was recorded. Number of subjects who developed or resolved lithiasis and developed or resolved sludge, comparing Baseline to V11 and to LVA are presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: The Safety population was defined as all subjects who received at least one dose of each IMP during the co-administration period (i.e. one dose of lanreotide Autogel 120 mg and one dose of pegvisomant).
Measure: Number; unit: participants
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
participants
  Developed Sludge: V11 vs V3 | 3
  Resolved Sludge: V11 vs V3 | 5
  Developed Lithiasis: V11 vs V3 | 1
  Resolved Lithiasis: V11 vs V3 | 1
  Developed Sludge: LVA vs V3 | 3
  Resolved Sludge: LVA vs V3 | 5
  Developed Lithiasis: LVA vs V3 | 2
  Resolved Lithiasis: LVA vs V3 | 1

21. Secondary Outcome: Change From Baseline in Mean Pituitary Tumour Size During the Co-administration Period
Description: Pituitary tumour size was assessed by Magnetic Resonance Imaging at V2, V3 and V11 (or in case of premature study discontinuation, at the early withdrawal visit). The two longest diameters of the pituitary tumour were to be measured. The change in mean pituitary tumour size from Baseline to V11 and to LVA is presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 53
mm^3
  Change at V11: number analyzed (Participants) | 49
  Change at V11 | 2.4 (729.7)
  Change at LVA | 6.3 (707.6)

22. Secondary Outcome: Change From Baseline in Mean Blood Glucose Maximum Concentration (Cmax) From Oral Glucose Tolerance Test (OGTT) During the Co-administration Period; Assessed in Non Diabetic Subjects
Description: Glucose tolerance was only evaluated in non diabetic subjects. Glucose tolerance was assessed based on measurement of fasting blood glucose and insulin levels taken at V2 and OGTT performed at V3 and V11 (or in case of premature study discontinuation, at the early withdrawal visit). A dose of 75 g oral glucose was given to subjects and blood samples then taken at 30, 60, 90 and 120 minutes after oral glucose to measure glucose, insulin and GH levels, and to evaluate the GH nadir level. The OGTT was performed after the assessment of IGF-1 and all safety laboratory tests, but before IMPs administration at V3. Glucose, insulin and GH levels were assessed before OGTT in fasting conditions and at the same time as IGF-1 assessment. The change in mean blood glucose Cmax (as determined from OGTT) from Baseline to V11 and to LVA is presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: The Safety population was defined as all subjects who received at least one dose of each IMP during the co-administration period (i.e. one dose of lanreotide Autogel 120 mg and one dose of pegvisomant). Assessed in non diabetic subjects only (n = 38). Only evaluable subjects with an assessment at the specified visit were included in the analysis.
Measure: Mean (Standard Deviation); unit: millimoles per litre (mmol/L)
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 38
millimoles per litre (mmol/L)
  Change at V11: number analyzed (Participants) | 34
  Change at V11 | 0.53 (1.72)
  Change at LVA | 0.61 (1.69)

23. Secondary Outcome: Change From Baseline in Mean Fasting Insulin Concentration During the Co-administration Period; Assessed in Non Diabetic Subjects
Description: Glucose tolerance was only evaluated in non diabetic subjects. Glucose tolerance was assessed based on measurement of fasting blood glucose and insulin levels taken at V2 and OGTT performed at V3 and V11 (or in case of premature study discontinuation, at the early withdrawal visit). A dose of 75 g oral glucose was given to subjects and blood samples then taken at 30, 60, 90 and 120 minutes after oral glucose to measure glucose, insulin and GH levels, and to evaluate the GH nadir level. The OGTT was performed after the assessment of IGF-1 and all safety laboratory tests, but before IMPs administration at V3. Glucose, insulin and GH levels were assessed before OGTT in fasting conditions and at the same time as IGF-1 assessment. The change in mean fasting insulin concentration from Baseline to V11 and to LVA is presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: picomoles per litre (pmol/L)
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 36
picomoles per litre (pmol/L)
  Change at V11: number analyzed (Participants) | 32
  Change at V11 | -12.7 (41.5)
  Change at LVA | -11.7 (40.8)

24. Secondary Outcome: Change From Baseline in Mean Fasting Glucose Concentration During the Co-administration Period; Assessed in Non Diabetic Subjects
Description: Glucose tolerance was only evaluated in non diabetic subjects. Glucose tolerance was assessed based on measurement of fasting blood glucose and insulin levels taken at V2 and OGTT performed at V3 and V11 (or in case of premature study discontinuation, at the early withdrawal visit). A dose of 75 g oral glucose was given to subjects and blood samples then taken at 30, 60, 90 and 120 minutes after oral glucose to measure glucose, insulin and GH levels, and to evaluate the GH nadir level. The OGTT was performed after the assessment of IGF-1 and all safety laboratory tests, but before IMPs administration at V3. Glucose, insulin and GH levels were assessed before OGTT in fasting conditions and at the same time as IGF-1 assessment. The change in mean fasting glucose concentration from Baseline to V11 and to LVA is presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 36
mmol/L
  Change at V11: number analyzed (Participants) | 32
  Change at V11 | -0.05 (0.71)
  Change at LVA | -0.09 (0.69)

25. Secondary Outcome: Change From Baseline in Mean Fasting Insulin / Glucose Ratio During the Co-administration Period; Assessed in Non Diabetic Subjects
Description: Glucose tolerance was only evaluated in non diabetic subjects. Glucose tolerance was assessed based on measurement of fasting blood glucose and insulin levels taken at V2 and OGTT performed at V3 and V11 (or in case of premature study discontinuation, at the early withdrawal visit). A dose of 75 g oral glucose was given to subjects and blood samples then taken at 30, 60, 90 and 120 minutes after oral glucose to measure glucose, insulin and GH levels, and to evaluate the GH nadir level. The OGTT was performed after the assessment of IGF-1 and all safety laboratory tests, but before IMPs administration at V3. Glucose, insulin and GH levels were assessed before OGTT in fasting conditions and at the same time as IGF-1 assessment. The change in mean fasting insulin / glucose ratio from Baseline to V11 and to LVA is presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 34
ratio
  Change at V11: number analyzed (Participants) | 30
  Change at V11 | -2.61 (8.12)
  Change at LVA | -2.33 (7.94)

26. Secondary Outcome: Change From Baseline in Mean Glycosylated Haemoglobin (HbA1C) During the Co-administration Period; Assessed in Non Diabetic and Diabetic Subjects
Description: Glycosylated haemoglobin (HbA1C) was measured at V2, V3 and V11 (or in case of premature discontinuation, at the early withdrawal visit). The change in mean HbA1C in diabetic and non diabetic subjects from Baseline to V11 and to LVA are presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: The Safety population was defined as all subjects who received at least one dose of each IMP during the co-administration period (i.e. one dose of lanreotide Autogel 120 mg and one dose of pegvisomant). Only evaluable subjects with an assessment at the specified visit were included in the analysis (56 overall for diabetic + non-diabetic subjects).
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 56
percentage
  Diabetic Subjects: Change at V11: number analyzed (Participants) | 18
  Diabetic Subjects: Change at V11 | -0.05 (0.71)
  Diabetic Subjects: Change at LVA: number analyzed (Participants) | 19
  Diabetic Subjects: Change at LVA | -0.05 (0.69)
  Non Diabetic Subjects: Change at V11: number analyzed (Participants) | 33
  Non Diabetic Subjects: Change at V11 | 0.05 (0.20)
  Non Diabetic Subjects: Change at LVA: number analyzed (Participants) | 37
  Non Diabetic Subjects: Change at LVA | 0.05 (0.21)

27. Secondary Outcome: Change From Baseline in Liver Function Test Parameters During the Co-administration Period
Description: Blood samples for clinical laboratory tests were taken at V1, V2, V3 and V11 (or in case of premature study discontinuation, at the early withdrawal visit). During the co-administration period, hepatic toxicity was assessed at each visit (V5 to V10) by measuring alanine amino transferase (ALT), aspartate amino transferase (AST), alkaline phosphatase, gamma glutamyl transferase (GGT), prothrombin time and total bilirubin. The change in mean ALT, AST, GGT and alkaline phosphatase from Baseline to V11 and to LVA are presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
IU/L
  AST: Change at V11: number analyzed (Participants) | 52
  AST: Change at V11 | 3.3 (10.7)
  AST: Change at LVA | 4.5 (13.0)
  ALT: Change at V11: number analyzed (Participants) | 52
  ALT: Change at V11 | 4.1 (11.7)
  ALT: Change at LVA | 7.8 (23.2)
  GGT: Change at V11: number analyzed (Participants) | 52
  GGT: Change at V11 | -1.0 (17.8)
  GGT: Change at LVA | 1.5 (20.8)
  Alkaline Phosphatase: Change at V11: number analyzed (Participants) | 52
  Alkaline Phosphatase: Change at V11 | -1.7 (14.5)
  Alkaline Phosphatase: Change at LVA | -0.8 (15.4)

28. Secondary Outcome: Change From Baseline in Total Bilirubin During the Co-administration Period
Description: Blood samples for clinical laboratory tests were taken at V1, V2, V3 and V11 (or in case of premature study discontinuation, at the early withdrawal visit). During the co-administration period, hepatic toxicity was assessed at each visit (V5 to V10) by measuring ALT, AST, alkaline phosphatase, GGT, prothrombin time and total bilirubin. The change in mean total bilirubin from Baseline to V11 and to LVA is presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: micromoles per litre
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
micromoles per litre
  Change at V11: number analyzed (Participants) | 52
  Change at V11 | -1.3 (2.9)
  Change at LVA | -1.2 (2.8)

29. Secondary Outcome: Change From Baseline in Prothrombin Time (Expressed as a Percentage of Normal) During the Co-administration Period
Description: Blood samples for clinical laboratory tests were taken at V1, V2, V3 and V11 (or in case of premature study discontinuation, at the early withdrawal visit). During the co-administration period, hepatic toxicity was assessed at each visit (V5 to V10) by measuring ALT, AST, alkaline phosphatase, GGT, prothrombin time and total bilirubin. Prothrombin time was expressed as a percentage of the time taken for a control blood sample to clot (designated as 100%) and the mean change from Baseline to V11 and to LVA is presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
percentage of time
  Change at V11: number analyzed (Participants) | 51
  Change at V11 | -3.7 (16.0)
  Change at LVA | -3.6 (15.2)

30. Secondary Outcome: Number of Subjects With Putative Antibodies to Lanreotide and to Pegvisomant During the Co-administration Period
Description: Presence of putative antibodies to lanreotide and antibodies to pegvisomant were assessed prior to IMP administration at V2, V4 and V11 (or in case of premature study discontinuation, at the early withdrawal visit). The number of subjects with putative antibodies to lanreotide and to pegvisomant during the co-administration period (Baseline up to V11) is presented.
Time Frame: V3 (Week 12; Baseline) up to V11 (Week 44)
Population: as for outcome 20
Measure: Number; unit: Number of subjects
Arm/Group | Lanreotide Autogel + Pegvisomant Co-administration
Number analyzed (Participants) | 57
Number of subjects
  Antibodies for Lanreotide | 4
  Antibodies for Pegvisomant | 6

ADVERSE EVENTS:
Time Frame: Run-in Period: approximately 16 weeks and Co-administration Period: approximately 28 weeks.
Description: Adverse event (AE) data is reported as treatment-emergent AEs for both the run-in and co-administration periods and is presented for the Safety Population, defined as all subjects who received at least one dose of each IMP (i.e. one dose of lanreotide Autogel 120 mg and one dose of pegvisomant during the co-administration period).
Groups:
- Run-in Period: During the 16 week run-in period, eligible subjects received one injection of lanreotide Autogel 120 mg every 28 days, administered by deep s.c. injection.
- Co-administration Period: During the 28 week co-administration period, eligible subjects received both lanreotide Autogel and pegvisomant concomitantly. The lanreotide Autogel dose during the co-administration period was fixed at 120 mg. Pegvisomant was administered once or twice a week via s.c. injection and the dose of could be adapted every 8 weeks based on IGF-1 levels, following a starting dose of 60 mg once a week (dose could vary from 40 to 120 mg per week and maximum permitted dose was 60 mg twice a week).
Arm/Group | Run-in Period | Co-administration Period
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 2/57 | 8/57
Other Adverse Events (participants affected / at risk) | 30/57 | 41/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Period (N=57) | Co-administration Period (N=57)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Facial palsy (Nervous system disorders) | 0 (0) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Period (N=57) | Co-administration Period (N=57)
Injection site nodule (General disorders) | 1 (1) | 2 (2)
Injection site pain (General disorders) | 2 (2) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 2 (4)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 5 (12) | 4 (7)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2)
Cytolytic hepatitis (Hepatobiliary disorders) | 0 (0) | 4 (4)
Cholelithiasis (Hepatobiliary disorders) | 6 (7) | 2 (3)
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 4 (4)
Nasopharyngitis (Infections and infestations) | 2 (2) | 5 (6)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No